CLINICAL TRIAL: NCT01028885
Title: A Prospective Study Implementing MRI Based Treatment Planning for Clinical Target Volume Definition and Immobilization in Post-Prostatectomy Radiation Treatment
Brief Title: MRI-Guided Radiation Therapy in Treating Patients Who Have Undergone Surgery to Remove the Prostate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 10809; NCI-2009-01441; NCT00977743 (obsolete NCT alias)
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Prostate Cancer; Adenocarcinoma of the Prostate; Stage I Prostate Cancer; Stage II Prostate Cancer; Stage III Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Radiotherapy, Image-Guided; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients undergo MRI and CT scan-based simulation for treatment planning with endorectal balloon target immobilization. The treatment target volumes and surrounding organs at risk are contoured, treatment plan developed and approved.
  Patients then undergo 39 fractions of image-guided intensity-modulated radiotherapy over 8 weeks. Patients also undergo weekly MRI scans of the pelvis (in the planned treatment position) during radiotherapy.
  Interventions: Procedure: radiation therapy treatment planning/simulation; Procedure: intensity-modulated radiation therapy; Procedure: image-guided radiation therapy; Procedure: magnetic resonance imaging; Procedure: computed tomography

INTERVENTIONS:
Procedure: radiation therapy treatment planning/simulation
Procedure: intensity-modulated radiation therapy
  Other Names: IMRT
Procedure: image-guided radiation therapy
Procedure: magnetic resonance imaging
  Other Names: MRI; NMR imaging; NMRI; nuclear magnetic resonance imaging
Procedure: computed tomography
  Other Names: tomography, computed

SUMMARY:
This is a prospective clinical trial examining the use of MRI to measure internal organ motion and any resulting changes in the target volume (shape and location) during a course of post-operative radiation therapy for prostate cancer. The goal is to better understand and characterize these physiologic variations so that they can be accounted for during the treatment planning process. The ultimate longer-term clinical goal here is to provide a form of adaptive radiation therapy in the future, such that if major changes are seen over an 8-week course of radiation therapy in our study. This may argue for hypofractionating those patients who are most likely to have major shifts over time.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the use of MRI in delineating clinical target volumes, as well as endorectal balloon target immobilization in patients treated with radiation following radical prostatectomy.

SECONDARY OBJECTIVES:

II. Trends over time in CTV, bladder and rectum volumes and percent change from baseline at each time point. III. Frequency of events in which the CTV falls outside the PTV. IV. Proportion of the total CTV which falls outside the PTV at each event. V. Trends over time in dose-volume exposures for bladder and rectum.

OUTLINE: Patients undergo MRI and CT scan-based simulation for treatment planning with endorectal balloon target immobilization. The treatment target volumes and surrounding organs at risk are contoured, treatment plan developed and approved.

Patients then undergo 39 fractions of image-guided intensity-modulated radiotherapy over 8 weeks. Patients also undergo weekly MRI scans of the pelvis (in the planned treatment position) during radiotherapy.

ELIGIBILITY:
Inclusion

* Completion of a radical prostatectomy for adenocarcinoma of the prostate
* Scheduled post-operative radiation therapy as part of the patient's treatment for prostate cancer
* Subjects are capable of giving informed consent

Exclusion

* The presence of grossly visualized or palpable disease recurrence
* Patients who are unable to undergo an MRI scan such as those with an implanted permanent pacemaker or ICD
* Patients with metastatic disease or an increasing PSA

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-06; Primary Completion 2012-02 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Clinical treatment target motion and deformation as quantified by co-registration of weekly MRI scans with original treatment planning MRI scans
Avoidance of any unexpected grade 3 or 4 toxicities

SECONDARY OUTCOMES:
Comparison of MRI and CT delineated target volumes defined during the treatment planning process
Distributions of clinical target volume (CTV), bladder and rectum volumes, and percent change from baseline
Incidence of CTV falling outside the planned treatment volume (PTV)
Distributions of the proportion of the total CTV which falls outside the PTV
Dose-volume exposures

CONTACTS AND LOCATIONS:
Overall Officials: Neha Vapiwala, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania, United States